CLINICAL TRIAL: NCT00402727
Title: A Prospective, Randomized, Double Dummy, Double Blind, Multinational, Multicenter Trial Comparing the Safety and Efficacy of Sequential (Intravenous/Oral) Moxifloxacin 400 mg OD to Intravenous Piperacillin/Tazobactam 4.0/0.5 g Every 8 Hours Followed by Oral Amoxicillin/Clavulanic Acid Tablets 875/125 mg Every 12 Hours for the Treatment of Subjects With Complicated Skin and Skin Structure Infections
Brief Title: Comparison of Sequential IV/PO Moxifloxacin With IV Piperacillin/Tazobactam Followed by PO Amoxicillin/Clavulanic Acid in Patients With a Complicated Skin and Skin Structure Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11974; 2006-001599-18 (EudraCT Number)
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Abscess; Wound Infection; Diabetic Foot; Ulcer
MeSH Terms: conditions — Abscess; Wound Infection; Diabetic Foot; Ulcer | interventions — Moxifloxacin; Piperacillin; Tazobactam; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Experimental): Moxifloxacin (Avelox, BAY 12-8039) 400 mg intravenous (IV) once daily followed by Moxifloxacin 400 mg oral tablets once daily for a minimum of 7 days and a maximum of 21 days. Oral phase was not always mandatory.
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- PIP/TAZ-AMC (Active Comparator): Piperacillin/Tacobactam 4.0/0.5 g (PIP/TAZ) administered intravenous three times daily followed by Amoxicillin/Clavulanic acid (AMC) oral tablets 875/125 mg twice daily for a minimum of 7 days and a maximum of 21 days. Oral phase not always mandatory.
  Interventions: Drug: Piperacillin/Tazobactam & Amoxicillin/Clavulanic acid

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Moxifloxacin (Avelox, BAY 12-8039) 400 mg intravenous (IV) once daily followed by Moxifloxacin 400 mg oral tablets once daily for a minimum of 7 days and a maximum of 21 days. Oral phase was not always mandatory.
  Arms: Moxifloxacin
Drug: Piperacillin/Tazobactam & Amoxicillin/Clavulanic acid — Piperacillin/Tacobactam 4.0/0.5 g (PIP/TAZ) administered intravenous three times daily followed by Amoxicillin/Clavulanic acid (AMC) oral tablets 875/125 mg twice daily for a minimum of 7 days and a maximum of 21 days. Oral phase not always mandatory.
  Arms: PIP/TAZ-AMC

SUMMARY:
Patients, who are considered suitable by their physicians to take part in this research, will have a physical examination (including an Electrocardiogram (ECG)), blood and urine samples taken, as well as a sample of the secretions or tissue around their infection site. In addition, the site of the infection will be photographed. The patients will be randomly assigned one of the treatments: intravenous (IV)/per oral (PO) moxifloxacin (drug under evaluation) or IV piperacillin/tazobactam followed by PO amoxicillin/clavulanic acid (i.e., one of the reference treatments for this kind of infection). The maximum treatment duration will be 21 days, and the minimum will be 7 days. During the hospitalization, the patients will have a physical examination every day. On Day 3-5 during therapy as well as at the end of treatment, the patients will have repeated examinations. These tests and evaluations will be repeated 14 to 28 days after the end of treatment. During this visit, blood and urine samples will be taken only if judged necessary by the physicians.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men or women of 18 years and above with a diagnosis of bacterial skin and skin structure infection that requires

  * Hospitalization and
  * Initial parenteral therapy for at least 48 hours and
  * Meets at least one of the following criteria:

    * Involvement of deep soft tissue (e.g. fascial, muscle layers)
    * Requirement for a significant surgical intervention including surgical drainage, drainage procedure guided by imaging and/or debridement
    * Association with a significant underlying disease that may complicate response to treatment. An underlying disease is considered significant if it includes any of the following conditions that are present at the time of presentation: cancer (except basal- or squamous-cell cancer of the skin), cardiac (i.e., congestive heart disease), diabetes mellitus, hepatic (i.e., cirrhosis or another form of chronic liver disease), immunologic, renal disease, respiratory, transplantation or vascular disease
* Duration of infection < 21 days
* Diagnosis of one of the following skin and skin structure infections that requires hospitalization and initial parenteral antibiotic therapy for at least 48 hours:

  * Major abscess(es) associated with extensive cellulitis, which requires antibiotic therapy in addition to surgical incision and drainage
  * Diabetic foot infection of mild to severe intensity (perfusion, extent/size, depth/tissue loss, infection and sensation (PEDIS) grade 2-4) in the presence or absence of osteomyelitis. Subjects with osteomyelitis may only be enrolled if the infected bone is completely removed by surgery and if residual infection requiring antibiotics is still present following surgery
  * Wound infection including: post surgical (surgical incision), post-traumatic, human bite/clenched fist and animal bite wound and wound associated with injection drug abuse:

    * Infections must have occurred within 30 days of a surgical procedure, trauma, animal bite, or human bite, and involve the skin and skin structures at the site of the incision, trauma, or bite
    * In addition, post-surgical/trauma wound infections must meet the following criteria:

      * Involvement of deep soft tissues (e.g. fascial and muscle layers) of the incision/trauma
      * At least one of the following criteria:

        * Purulent drainage from the deep incision/trauma
        * Identification of an infecting organism from an aseptically obtained culture of fluid or tissue from incision/trauma
      * At least one of the following signs and symptoms:

        * Localized pain or tenderness
        * Fever (see below) AND the incision (in case of post-surgical wound infections) is deliberately opened by a surgeon, unless the culture is negative
        * Abscess or other evidence of infection involving the deep incision/trauma, found on direct examination, during reoperation/operation (in case of trauma), or by histologic or radiologic examination
      * Diagnosis of a deep incisional/post-trauma Skin Structure Infections (SSI) by a surgeon or attending physician
      * Bite wounds/clenched fist infections and wounds associated with injection drug abuse must meet the criteria defining a Complicated Skin and Skin Structure Infections (cSSSI)
  * Infected ischemic ulcers with at least one of the following conditions:

    * Peripheral vascular disease
    * Conditions pre-disposing to pressure sores such as paraplegia, peripheral neuropathy
    * Presence of at least 3 of the following signs or symptoms:

      * Purulent drainage or discharge
      * Erythema extending > 1 cm from the wound edge
      * Fluctuance
      * Pain or tenderness to palpation
      * Swelling or induration
      * Fever, defined as body temperature

        * > 37.5°C (axillary)
        * > 38°C (orally)
        * > 38.5°C (tympanically) or
        * > 39°C (rectally)

          * OR
        * Elevated total peripheral white blood cell (WBC) count > 12,000/mm3 or
        * >15 % immature neutrophils (bands) regardless of total peripheral WBC count
      * C reactive protein (CRP) >20 mg/L
* Specimen obtained for culture from infected area by needle aspiration of obviously purulent material or by tissue biopsy or by curettage of the surface of ulcer within 48 hours prior to the initiation of study drug therapy
* Duration of treatment of the skin/skin structure infection is anticipated to be at least 7 days.
* Surgical drainage or debridement of infected wounds or abscesses, if necessary, have to have been completed <= 48 hours after the initiation of study drug therapy

Exclusion Criteria:

* Women, who are pregnant or lactating, or in whom pregnancy can not be excluded (Note: a urine pregnancy test has to be performed for all women of childbearing potential before randomization to the study drug)
* The following skin and skin structure infections:

  * Necrotizing fasciitis including Fourniers gangrene, ecthyma gangrenosum, streptococcal necrotizing fasciitis and clostridial necrotizing fasciitis
  * Burn wound infections
  * Secondary infections of a chronic skin disease (e.g. atopic dermatitis)
  * Infection of prosthetic materials (e.g. subcutaneous tissue infection related to a central venous catheter or permanent cardiac pacemaker battery pack). Subjects with removal of a prosthetic device involved in an infection should not be included
  * Infections where a surgical procedure alone is definitive therapy
  * Subjects with uncomplicated skin and skin structure infections including folliculitis and furunculosis, carbunculosis, simple abscesses and superficial cellulitis
* Known hypersensitivity to quinolones and/or any type of beta-lactam antibiotic drugs or any of the excipients
* Previous history of cholestatic jaundice/hepatic dysfunction associated with amoxicillin-clavulanic acid
* Severe, life threatening disease with a life expectancy of less than 2 months
* Immunosuppression including:

  * Known neutropenia (neutrophil count < 1000/µL)
  * Known lymphopenia with absolute CD4+ T cell count < 200/mm3
  * Acquired immunodeficiency syndrome (AIDS)-defining event and/or concomitant therapy with Highly Active Antiretroviral Therapy (HAART)
  * Chronic treatment (>/= 2 weeks) with known immunosuppressant therapy (including treatment with > 15 mg/day of systemic prednisone or equivalent)
  * Any other congenital or acquired immune defect or immunosuppression
* Known severe hepatic insufficiency (Child Pugh C) or transaminases increase > 5 fold upper limit of normal (ULN)
* Known renal impairment with a baseline measured or calculated serum creatinine clearance < 40 mL/min
* Known prolongation of the QT interval or concomitant use of drugs reported to increase the QT interval (e.g. Class IA or Class III antiarrhythmics [eg., quinidine, procainamide, amiodarone, sotalol], neuroleptics [e.g. haloperidol], tricyclic antidepressive agents, certain antimicrobials [e.g. pentamidine, halofantrine], certain antihistaminics [e.g. terfenadine], and other [cisapride, vincamine IV, depridil, diphemanil])
* Uncorrected hypokalemia
* Clinically relevant bradycardia
* Clinically relevant heart failure with reduced left ventricular ejection fraction (i.e., below 40%)
* Previous history of symptomatic arrhythmias
* Previous history of tendon disease/disorder with quinolones
* Known or suspected concomitant bacterial infection requiring additional systemic antibacterial treatment, e.g. underlying septic arthritis
* Requiring therapy with probenecid
* Treatment with a systemic or topical antibacterial agent for > 24 hours in the previous 7 days preceding study entry unless the subject showed no response or had worsening of clinical signs and symptoms despite 3 or more days of prior therapy and a culture obtained at the time of subject enrollment showed persistence of a pathogen which is susceptible to the study drugs. The prior antimicrobial therapy must not have been a fluoroquinolone or a beta lactam/beta lactamase combination
* Infection known to be due to a Methicillin-Resistant Staphylococcus Aureus (MRSA), Methicillin-Resistant Staphylococcus Epidermidis (MRSE) or Vancomycin Resistant Enterococcus (VRE) as the single isolated pathogen
* Previous enrolment in this study
* Participation in any clinical investigational drug study within 4 weeks of screening
* Previous history of seizure disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (98):
- Austria (3):
  - Graz, Styria
  - Graz
  - Vienna
- Belgium (3):
  - Bornem
  - Bruxelles - Brussel
  - Edegem
- Bulgaria (4):
  - Dobrich
  - Pleven
  - Rousse
  - Sofia
- France (9):
  - Annecy
  - Avignon
  - Boulogne-sur-Mer
  - Denain
  - Grenoble
  - Le Grau-du-Roi
  - Nevers
  - Quimper
  - Tourcoing
- Germany (11):
  - Mannheim, Baden-Wurttemberg
  - München, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Wiesbaden, Hesse
  - Hanover, Lower Saxony
  - Bochum, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Magdeburg, Saxony-Anhalt
  - Lübeck, Schleswig-Holstein
- Greece (5):
  - Athens, Attica
  - Athens, Greece
  - Athens
  - Rio Patras
  - Thessaloniki
- Hungary (6):
  - Budapest
  - Debrecen
  - Győr
  - Kaposvár
  - Székesfehérvár
  - Veszprém
- Ireland (5):
  - Wilton, Cork
  - Dublin, Dublin
  - Galway, Galway
  - Dublin
  - Sligo
- Israel (2):
  - Haifa
  - Tel Litwinsky
- Italy (5):
  - Chieti
  - Milan
  - Pavia
  - Roma
  - Siena
- Latvia (4):
  - Daugavpils
  - Liepāja
  - Riga
  - Valmiera
- Lithuania (4):
  - Kaunas
  - Šiauliai
  - Ukmerge
  - Vilnius
- Netherlands (2):
  - Alkmaar
  - Eindhoven
- Poland (5):
  - Krakow
  - Lublin
  - Poznan
  - Puławy
  - Warsaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iași
- Russia (4):
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Yaroslavl
- South Africa (4):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Cape Town, Western Cape
  - Worcester, Western Cape
- Spain (5):
  - Barcelona, Barcelona
  - Terrassa (Barcelona), Catalonia
  - Madrid, Madrid
  - Oviedo, Principality of Asturias
  - Salamanca, Salamanca
- Ukraine (5):
  - Ivano-Frankivsk
  - Kiev
  - Lviv
  - Odesa
  - Uzhhorod
- United Kingdom (9):
  - London, Greater london
  - Winchester, Hampshire
  - Inverness, Highland
  - Edinburgh, Lothian
  - Manchester, Manchester
  - Glasgow, Stratchclyde
  - Newcastle upon Tyne, Tyne and Wear
  - Leeds, West Yorkshire
  - York, York

REFERENCES:
- [Result] Gyssens IC, Dryden M, Kujath P, Nathwani D, Schaper N, Hampel B, Reimnitz P, Alder J, Arvis P. A randomized trial of the efficacy and safety of sequential intravenous/oral moxifloxacin monotherapy versus intravenous piperacillin/tazobactam followed by oral amoxicillin/clavulanate for complicated skin and skin structure infections. J Antimicrob Chemother. 2011 Nov;66(11):2632-42. doi: 10.1093/jac/dkr344. Epub 2011 Sep 6. PMID 21896561
- [Result] Schaper NC, Dryden M, Kujath P, Nathwani D, Arvis P, Reimnitz P, Alder J, Gyssens IC. Efficacy and safety of IV/PO moxifloxacin and IV piperacillin/tazobactam followed by PO amoxicillin/clavulanic acid in the treatment of diabetic foot infections: results of the RELIEF study. Infection. 2013 Feb;41(1):175-86. doi: 10.1007/s15010-012-0367-x. Epub 2012 Nov 23. PMID 23180507
- [Derived] D'Onofrio V, Monnier AA, Kremer C, Stappers MHT, Netea MG, Gyssens IC. Lesion size is associated with genetic polymorphisms in TLR1, TLR6, and TIRAP genes in patients with major abscesses and diabetic foot infections. Eur J Clin Microbiol Infect Dis. 2020 Feb;39(2):353-360. doi: 10.1007/s10096-019-03732-7. Epub 2019 Nov 30. PMID 31786695
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 834 subjects with complicated skin and skin structure infections (cSSSI) enrolled based on evaluation (by interview, medical history, physical examination, and laboratory tests); 21 subjects not randomized, 668 subjects (361 on moxifloxacin, 307 on pipercillin/tazobactam plus amoxicillin/clavulanic acid) included in primary efficacy analysis.
Period: Overall Study
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Started | 432 | 381
Achieving End Of Treatment (EOT) | 408 | 355
Achieving Test Of Cure (TOC) | 390 | 347
Completed | 390 | 347
Not Completed | 42 | 34
Not completed — Adverse Event | 10 | 6
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 24 | 11
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 3 | 7
Not completed — supply problems | 2 | 1
Not completed — non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin | PIP/TAZ-AMC | Total
Number analyzed (Participants) | 432 | 381 | 813
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (16) | 54 (16) | 53 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 123 | 284
  Male | 271 | 258 | 529
Primary diagnosis [Number; unit: Participants]
  Major abscess | 184 | 170 | 354
  Diabetic foot infection | 123 | 110 | 233
  Wound infection | 72 | 55 | 127
  Infected ischemic ulcer | 24 | 18 | 42
  No cSSSI | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cured Participants as Determined by the Data Review Committee (DRC) at Test of Cure Visit in the Per Protocol (PP) Population
Description: Clinical response was evaluated by the DRC and graded as "cure", "failure" or "indeterminate" at the TOC visit. Members of the DRC were provided with subject data from the study database that included clinical signs and symptoms at each visit, concomitant medication, microbiology results, laboratory tests and interpretation of photographs.
Time Frame: 14 - 28 days after last dose of study medication
Population: The per protocol population was the main analysis set for the assessment of clinical response and was defined as those subject with no major protocol deviations that would have influenced the primary outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 361 | 307
percentage of participants | 88.6 | 89.6
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; Calculated were 95% confidence intervals for the difference in success rates between treatment groups (moxifloxacin minus comparator). Method as described in Koch et al; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set to 10% in the protocol, in agreeance with FDA recommendations. Sample size was estimated using the method as described in Farrington-Manning. Estimation was performed to achieve 85% power, based on the equivalence delta of 10%, and a clinical success rate of 80% in the per protocol population; Difference of cure rates (in percent) = -1.0, 95% CI [-5.3 to 3.9] — A positive value indicates an advantage for the treatment group of moxifloxacin, a negative value an advantage for the comparator group

2. Secondary Outcome: Percentage of Cured Participants as Determined by the Data Review Committee (DRC) at Test of Cure Visit in the Intent to Treat (ITT) Population
Description: as for outcome 1
Time Frame: 14 - 28 days after last dose of study medication
Population: The intent-to-treat population was the analysis set used for the assessment of clinical response and was defined as all randomized subject that received at least one dose of study medication and had at least one observation after intake of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 426 | 377
percentage of participants | 82.2 | 80.9
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of cure rates (in percent) = 1.3, 95% CI [-3.8 to 6.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Assessed as Improvements by the Data Review Committee (DRC) at the During Treatment Day 3-5 in the Per Protocol (PP) Population
Description: Clinical response was evaluated by the investigator and graded as "improvement in signs and symptoms," or "failure to respond," or "indeterminate" at Day 3 to 5 after treatment start based on subject data for clinical signs and symptoms at each visit, concomitant medication, microbiology results, laboratory tests and interpretation of photographs.
Time Frame: 3 - 5 days after start of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 361 | 307
percentage of participants | 98.3 | 99.0
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of improvement rates (in %) = -0.7, 95% CI [-1.6 to 0.6] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Assessed as Improvements by the Data Review Committee (DRC) at the During Treatment Day 3-5 in the Intent to Treat (ITT) Population
Description: as for outcome 3
Time Frame: 3 - 5 days after start of treatment
Population: The intent-to-treat population was the analysis set used for the assessment of clinical response and was defined as those subject with no major protocol deviations that would have influenced the secondary outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 426 | 377
percentage of participants | 97.2 | 95.8
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of improvement rates (in %) = 1.4, 95% CI [-1.3 to 3.9] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Assessed as Resolution by the Data Review Committee (DRC) at End of Therapy in the Per Protocol (PP) Population
Description: Clinical response was evaluated by the investigator and graded as "resolution," or "failure to respond," or "indeterminate" at the end of therapy based on subject data for clinical signs and symptoms at each visit, concomitant medication, microbiology results, laboratory tests and interpretation of photographs.
Time Frame: after 7 - 21 days of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 361 | 307
percentage of participants | 95.3 | 95.1
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of resolution rates (in %) = 0.2, 95% CI [-3.1 to 2.4] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Assessed as Resolution by the Data Review Committee (DRC) at End of Therapy in the Intent to Treat (ITT) Population
Description: Clinical response was evaluated by the investigator and graded as "resolution", or "failure to respond," or "indeterminate" at the end of therapy based on subject data for clinical signs and symptoms at each visit, concomitant medication, microbiology results, laboratory tests and interpretation of photographs.
Time Frame: after 7 - 21 days of treatment
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 426 | 377
percentage of participants | 92.3 | 90.7
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of resolution rates (in %) = 1.6, 95% CI [-2.4 to 5.3] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants With Bacteriological Success (BS) at 3 to 5 Days After Start of Treatment in the ITT Population With Causative Organisms
Description: Bacteriological success was defined as presumed eradication or eradication without superinfection. Presumed eradication was defined as clinical cure in absence of a culture, eradication as a negative culture, superinfection as appearance of a new organism.
Time Frame: 3 - 5 days after start of treatment
Population: The ITT population with causative organism population included all ITT subjects with least one causative organism that could be cultured from an appropriate specimen within 48 hours prior to or following randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 313 | 290
percentage of participants | 54.6 | 63.1
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of eradication rates (in %) = -8.5, 95% CI [-17.0 to -1.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Participants With Bacteriological Success (BS) at 3 to 5 Days After Start of Treatment in the Microbiological Valid (MBV) Population
Description: as for outcome 7
Time Frame: 3 - 5 days after start of treatment
Population: Microbiologically valid subjects were defined as all valid PP subjects in whom at least one causative organism could be cultured from an appropriate specimen within 48 hours prior to or following randomization and where a bacteriological evaluation at TOC visit was available and different from "indeterminate".
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 268 | 243
percentage of participants | 55.2 | 63.8
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of eradication rates (in %) = -8.6, 95% CI [-17.6 to -0.4] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants With Bacteriological Success (BS) After 7 - 21 Days of Treatment in the ITT Population With Causative Organisms
Description: Bacteriological success is presumed eradication or eradication without recurrence or superinfection. Presumed eradication was defined as clinical cure in absence of a culture, eradication as a negative culture, recurrence as reappearance of organism present at start of study, superinfection as appearance of a new organism.
Time Frame: after 7 - 21 days of treatment
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 313 | 290
percentage of participants | 84.0 | 87.9
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of eradication rates (in %) = -3.9, 95% CI [-9.5 to 1.4] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percentage of Participants With Bacteriological Success (BS) After 7 - 21 Days of Treatment in the Microbiological Valid (MBV) Population
Description: as for outcome 9
Time Frame: after 7 - 21 days of treatment
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 230 | 222
percentage of participants | 85.8 | 91.4
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of eradication rates (in %) = -5.6, 95% CI [-11.4 to -0.8] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percentage of Participants With Bacteriological Success (BS) After 14 - 28 Days After Last Dose of Study Medication in the ITT Population With Causative Organisms
Description: BS is presumed eradication or eradication without recurrence, super- or reinfection. Presumed eradication was defined as clinical cure in absence of a culture, eradication as a negative culture, recurrence as reappearance of organism present at start of study; super-, reinfection as appearance of a new organism during/after treatment.
Time Frame: 14 - 28 days after last dose of study medication
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 313 | 290
percentage of participants | 78.9 | 79.0
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of eradication rates (in %) = -0.1, 95% CI [-6.9 to 5.4] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percentage of Participants With Bacteriological Success (BS) After 14 - 28 Days After Last Dose of Study Medication in the Microbiological Valid (MBV) Population
Description: as for outcome 11
Time Frame: 14 - 28 days after last dose of study medication
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Number analyzed (Participants) | 226 | 212
percentage of participants | 84.3 | 87.2
Statistical Analysis 1: Comparison: Moxifloxacin vs PIP/TAZ-AMC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of eradication rates (in %) = -2.9, 95% CI [-9.3 to 2.2] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Moxifloxacin | PIP/TAZ-AMC
Serious Adverse Events (participants affected / at risk) | 21/426 | 14/377
Other Adverse Events (participants affected / at risk) | 35/426 | 20/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin (N=426) | PIP/TAZ-AMC (N=377)
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Necrosis (General disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Diabetic gangrene (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 3
Localised infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 2 | 0
Muscle abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Suture insertion (Surgical and medical procedures) | 1 | 0
Skin implant (Surgical and medical procedures) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Lymphorrhoea (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin (N=426) | PIP/TAZ-AMC (N=377)
Diarrhoea (Gastrointestinal disorders) | 10 | 8
Nausea (Gastrointestinal disorders) | 5 | 3
Pyrexia (General disorders) | 7 | 3
Electrocardiogram QT prolonged (Investigations) | 1 | 5
Headache (Nervous system disorders) | 5 | 3
Hypertension (Vascular disorders) | 11 | 2

LIMITATIONS AND CAVEATS:
Ten patients (six from the moxifloxacin group and 4 from the comparator group) did not receive study medication. They were excluded from the safety analyses. No adverse events were reported in these patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Bayer informs coordinating investigator's hospital that such publication could be expected to have an adverse effect on the confidentiality of any confidential information, then the coordinatin investigator's hospital shall prevent the publication, unless the confidential information can be deleted from the publication without having adetrimental effect on the scientific correctness of the publication.